CLINICAL TRIAL: NCT04115683
Title: Effect of Dual Task Training on Balance, Gait, Cognition and Neurotrophic Factors in Parkinson's Disease
Brief Title: Dual Task Training in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Çağrı Gülşen, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14.01.2019/35
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Dual Task Training
- Control Group (Active Comparator)
  Interventions: Other: Single Task Training

INTERVENTIONS:
Other: Dual Task Training — 45 minutes of dual task training consisting of motor activities (walking, balance... etc.) with combination of cognitive activities (spelling words, image description, nomination, word generation, counting... etc.) at sime time.
  Arms: Intervention Group
Other: Single Task Training — 45 minutes of single task training consisting of same motor activities (walking, balance... etc.)
  Arms: Control Group

SUMMARY:
The aim of study is to analyze the effects of dual task training on balance, gait, cognition and neurotrophic factors in Parkinson's disease.

DETAILED DESCRIPTION:
20 patients diagnosed with Parkinson's disease will be randomly assigned to either intervention or control group. And 10 healty subjects will be included to study in order to determine the reference values.The intervention group will be recieved cognitive and motor dual task training consisting of balance and walking activities 3 days a week for 8 weeks. Control group will be recieved same balance and walking activities in single task condition 3 days a week for 8 weeks. In order to evaluate the effects of the training, evaluations will be performed before and after the training period.

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age
* neurologist-diagnosed Parkinson's Disease
* Hoehn & Yahr (H&Y) stages 1 to 3
* 24 or more mini mental status examination score.

Exclusion Criteria:

* other neurologic disorder
* cardiovascular, inflammatory,vestibular or musculoskeletal problems that could prevent them to participate in an exercise program
* had deep brain stimulation history
* visual, auditory, orientational problems that could affect study results

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Balance-Postural Stability | 8 weeks
  Postural Stability will be evaluated with Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York).. Postural Stability test will performed on both feet and on the left and right foot separately. Total stability index score will obtained as the test result.
Balance- Limits of Stability | 8 weeks
  Limits of Stability will be evaluated with Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). Limits of Stability test assesses how much the center of gravity is displaced on the support surface without losing balance during the standing position. Total direction control score will obtained as the test result.
Balance- Modified Sensory Organization Tests | 8 weeks
  Modified Sensory Organization Tests will be evaluated Biodex Biosway Portable Balance System (Biodex Medical Systems Inc., Shirley, New York). MSOT assesses the effects of somatosensory, visual and vestibular senses on postural control during the standing position. It evaluates the sensory component of balance in two different visual conditions and on two different support surfaces; condition 1: eyes open-firm surface, condition 2: eyes closed-firm surface, condition 3: eyes open-foam surface and condition 4: eyes closed-foam surface. Stability index scores will obtained as the test result.
Gait Speed | 8 weeks
  Gait speed will be evaluated by using the BTS-G Walk system and recorded as m/min. It is a wireless system positioned on L5 vertebrae of the spine. It allows a functional objective gait analysis to be performed.
Cadence | 8 weeks
  Cadence will be evaluated by using the BTS-G Walk system and recorded as strides/min. It is a wireless system positioned on L5 vertebrae of the spine. It allows a functional objective gait analysis to be performed.
Stride width | 8 weeks
  Stride width will be evaluated by using the BTS-G Walk system and recorded as meters. It is a wireless system positioned on L5 vertebrae of the spine. It allows a functional objective gait analysis to be performed.
Stride length | 8 weeks
  Stride length will be evaluated by using the BTS-G Walk system and recorded as meters. It is a wireless system positioned on L5 vertebrae of the spine. It allows a functional objective gait analysis to be performed.
Montreal Cognitive Assessment (MoCA) | 8 weeks
  Montreal Cognitive Assessment (MoCA) will be used in order to evaluate cognition. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.It' score ranged from 0 to 30 and higher points indicates better cognitive outcomes.
Change in brain derived neurotrophic factor (BDNF) levels of serum | 8 weeks
  Brain derived neurotrophic factor (BDNF) levels of serum will be measured by using sandwich enzyme-linked immunosorbent assay (ELISA) kit.
Change in vascular endothelial growth factor (VEGF) levels of serum | 8 weeks
  Vascular endothelial growth factor (VEGF) levels of serum will be measured by using sandwich enzyme-linked immunosorbent assay (ELISA) kit.
Change in insulin like growth factor 1 (IGF-1) levels of serum | 8 weeks
  Insulin like growth factor 1 (IGF-1) levels of serum will be measured by using sandwich enzyme-linked immunosorbent assay (ELISA) kit.

SECONDARY OUTCOMES:
Hoehn and Yahr Scale for level of physical disability in Parkinson's disease. | 8 weeks
  Hoehn and Yahr Scale is measures level of physical disability in Parkinson's disease and stages patients between level 1 level 5. Higher level indicates worse physical condition.
Unified Parkinson's Disease Rating Scale (UPDRS) | 8 weeks
  The Unified Parkinson's Disease Rating Scale (UPDRS) is a widely used measure of impairment and disability associated with Parkinson's Disease (PD) consisting of four sections: (1) Mentation, behavior, and mood; (2) Activities of daily living (ADLs); (3) Motor; and (4) Complications.Sections I through III are scored using a 5-point Likert-type scale (0 = no impairment; 4 = marked impairment). Although individual sections are scored and reported independently, scores from sections I through III are also summed to provide a UPDRS Total score. The UPDRS total score ranges between 0 and 199 points. Higher points indicates worse outcome.
Berg Balance Scale (BBS) | 8 weeks
  Berg Balance Scale (BBS) is a scale that using for assess postural stability. It ranges 0-56 with higher score indicates better stability.
One-legged Stance Test | 8 weeks
  The duration participant is able to maintain their balance on one leg up to will be recorded.
Timed Up and Go (TUG) test | 8 weeks
  Time in seconds a person needs to stand up from a chair, walk a distance of 3 meters, turn around a flag, come back and sit down again.
Activities-Specific Balance Confidence (ABC) Scale | 8 weeks
  Activities-specific Balance Confidence scale (ABC), to quantify the level of confidence in performing a specific task without losing balance or becoming unsteady.
Stroop Test | 8 weeks
  Stroop test will be used to test cognitive function.
Trail Making Test (TMT) Part A and B | 8 weeks
  The Trail Making Test is a measure of attention, speed and mental flexibility.
Short-Form 8-Item Parkinson's Disease Questionnaire (PDQ-8) | 8 weeks
  The short-form 8-item Parkinson's disease Questionnaire (PDQ-8) is the most commonly used scale measuring health related quality of life (HRQoL) in PD patients. It includes 8 items, and each item has five options (never, occasionally, sometimes, often, always or cannot do at all). The total score ranges from 0 to 32. Higher scores indicates poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No